CLINICAL TRIAL: NCT00003883
Title: A Randomized, Comparative Study of Itraconazole Versus Fluconazole for Prevention of Aspergillus Infections in Peripheral Blood Stem Cell and Marrow Transplant Recipients
Brief Title: Itraconazole Compared With Fluconazole to Prevent Infections in Patients Undergoing Peripheral Stem Cell or Bone Marrow Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 1322.00; FHCRC-1322.00; NCI-H99-0030; CDR0000067050 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; chronic idiopathic myelofibrosis; childhood acute promyelocytic leukemia (M3); testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent ovarian germ cell tumor; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; infection; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; previously treated childhood rhabdomyosarcoma; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Infections; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Fluconazole; Itraconazole

INTERVENTIONS:
Drug: fluconazole
Drug: itraconazole

SUMMARY:
RATIONALE: Giving itraconazole or fluconazole may be effective in preventing infections in patients undergoing peripheral stem cell or bone marrow transplantation. It is not yet known whether itraconazole is more effective than fluconazole for preventing infections.

PURPOSE: Randomized phase III trial to compare the effectiveness of itraconazole with fluconazole to prevent infections in patients undergoing peripheral stem cell or bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of itraconazole versus fluconazole in reducing the incidence of breakthrough Aspergillus infections in patients undergoing allogeneic peripheral blood stem cell or bone marrow transplantation. II. Compare the incidence of combined mold/yeast infections and the use of alternative systemic antifungal treatments in these patients on this regimen. III. Compare the toxic effects of these two drugs in these patients. IV. Determine the survival rate of these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms. Arm I: Patients receive fluconazole orally or IV daily beginning at start of conditioning regimen and continuing until day 180 or until 4 weeks after stopping corticosteroids (if it occurs between days 120-180). Arm II: Patients receive oral fluconazole daily beginning at start of conditioning regimen and continuing until day 0. Patients then receive itraconazole orally or IV daily beginning on day 0 and continuing until day 180, or until 4 weeks after stopping corticosteroids (if it occurs between days 120-180).

PROJECTED ACCRUAL: A total of 578 patients (289 per arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Scheduled to undergo allogeneic peripheral blood stem cell, bone marrow, or cord blood transplant (except minitransplant) No documented or suspected invasive fungal infection

PATIENT CHARACTERISTICS: Age: 13 and over Performance status: Not specified Life expectancy: More than 2 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than 5 times upper limit of normal (ULN) OR AST or ALT no greater than 5 times ULN OR Alkaline phosphatase no greater than 5 times ULN Renal: Not specified Other: Weight at least 40 kg Fertile patients must use effective contraception No history of anaphylaxis due to azole antifungal drug compounds No uncontrolled bacteremia No concurrent condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No prior nonmyeloablative regimen (e.g., FHCRC-1209 or FHCRC-1225) No other concurrent antifungal agents No concurrent astemizole, terfenadine, or cisapride

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 1998-10; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren A. Marr, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington